CLINICAL TRIAL: NCT03716830
Title: Enhancing Acupuncture Treatment Effect Through Non-invasive Neuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Associate Professor, Associate Researcher, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2018P001970
Record Dates: First submitted 2018-10-18; First posted 2018-10-23 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of four groups: 1) verum acupuncture + real tDCS, 2) sham acupuncture + real tDCS, 3) verum acupuncture + sham tDCS, and 4) sham acupuncture + sham tDCS.
Who Masked: Participant, Investigator
Masking Description: Both participants and study staff will be blinded to the treatment group of participants. Only the licensed acupuncturist will be aware of the type of acupuncture the participant will be receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- verum acupuncture + real tDCS (Experimental)
  Interventions: Device: verum acupuncture; Device: real tDCS
- sham acupuncture + real tDCS (Experimental)
  Interventions: Device: sham acupuncture; Device: real tDCS
- verum acupuncture + sham tDCS (Experimental)
  Interventions: Device: verum acupuncture; Device: sham tDCS
- sham acupuncture + sham tDCS (Sham Comparator)
  Interventions: Device: sham acupuncture; Device: sham tDCS

INTERVENTIONS:
Device: verum acupuncture — Participants will receive real acupuncture treatment.
  Arms: verum acupuncture + real tDCS; verum acupuncture + sham tDCS
Device: sham acupuncture — Participants will receive sham acupuncture treatment.
  Arms: sham acupuncture + real tDCS; sham acupuncture + sham tDCS
Device: real tDCS — Participants will receive real transcranial direct current stimulation.
  Arms: sham acupuncture + real tDCS; verum acupuncture + real tDCS
Device: sham tDCS — Participants will receive sham transcranial direct current stimulation.
  Arms: sham acupuncture + sham tDCS; verum acupuncture + sham tDCS

SUMMARY:
In this study, investigators will examine the brain mechanism behind the synergistic effects of combining acupuncture and transcranial direct current stimulation (tDCS) treatments. Specifically, chronic low back pain (cLBP) patients will be recruited and randomized to one of four groups (30 per group, one month of treatment): 1) verum acupuncture + real tDCS, 2) sham acupuncture + real tDCS, 3) verum acupuncture + sham tDCS, and 4) sham acupuncture + sham tDCS. Investigators will study 1) the longitudinal (one-month) effects of different treatments as indicated by changes in resting state functional connectivity (rsFC), cerebral blood flow (CBF), clinical outcomes of low back pain, and quantitative sensory test (QST) and 2) the association between these changes.

ELIGIBILITY:
Inclusion Criteria:

* volunteers 18-60 years of age
* meet the classification criteria of chronic low back pain (having low back pain for more than 6 months), as determined by the referring physician
* at least 4/10 clinical pain on the 11-point Low Back Pain Numeric Rating Scale (LBP NRS)
* at least a 10th grade English-reading level; English can be a second language provided that the patients understand all questions used in the assessment measures

Exclusion Criteria:

* history of epilepsy or loss consciousness (LOC)
* specific causes of back pain (e.g. cancer, fractures, spinal stenosis, infections)
* complicated back problems (e.g. prior back surgery, medicolegal issues)
* the intent to undergo surgery during the time of involvement in the study
* history of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcomes. For example: asthma or claustrophobia
* presence of any contraindications to magnetic resonance imaging (MRI) scanning. For example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, inability to remain still in MRI scanner
* history of medical or psychiatric illness as determined by the investigator
* history of substance abuse or dependence

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started on Nov, 07, 2020. The study was conducted at Massachusetts General Hospital.
Period: Overall Study
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Started | 31 | 30 | 26 | 29
Completed | 27 | 25 | 20 | 23
Not Completed | 4 | 5 | 6 | 6
Not completed — Withdrawal by Subject | 2 | 2 | 6 | 5
Not completed — Adverse Event | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data analysis was performed based on group distribution.
Groups:
- Total: Total of all reporting groups
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS | Total
Number analyzed (Participants) | 27 | 25 | 20 | 23 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (13) | 38 (13) | 41 (13) | 42 (12) | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 10 | 11 | 48
  Male | 14 | 11 | 10 | 12 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 18 | 11 | 15 | 63
  Black or African | 4 | 2 | 4 | 2 | 12
  Asian | 2 | 5 | 2 | 2 | 11
  Other | 1 | 0 | 2 | 1 | 4
  Unknown/not-reported | 1 | 0 | 1 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 20 | 23 | 95

OUTCOME MEASURES:

1. Primary Outcome: Periaqueductal Gray (PAG) Resting State Functional Connectivity (rsFC) Changes
Description: We investigated whether tDCS and acupuncture treatments modulate resting-state functional connectivity (rsFC) of the periaqueductal gray (PAG). This was evaluated by comparing pre- and post-treatment MRI scans. In this report, we focused on the rsFC between the PAG and the rostral anterior cingulate cortex (rACC, peak MNI coordinate (2, 38, 12) with a 2-mm radius sphere). Functional connectivity values were computed as Pearson's correlation coefficients between the mean time series of predefined regions of interest (ROIs). To improve normality and enable parametric statistical analysis, these correlation coefficients (r) were converted to Fisher z values using the transformation z = 0.5 × ln[(1 + r) / (1 - r)]. Higher Fisher z values indicate stronger positive connectivity, whereas lower values indicate weaker or negative connectivity. Changes in Fisher z values from baseline to post-intervention reflect the degree and direction of connectivity modulation.
Time Frame: difference between Day 1 (pre-intervention); post-intervention at Week 4 (pre-intervention - Post-intervention)
Population: Individuals with chronic low back pain
Measure: Mean (Standard Deviation); unit: Fisher z-transformed correlation coeffic
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Number analyzed (Participants) | 24 | 23 | 19 | 21
Fisher z-transformed correlation coeffic | -0.03 (0.16) | 0.02 (0.17) | 0.11 (0.1) | -0.03 (0.11)

2. Secondary Outcome: Clinical Outcomes as Measured by LBP Intensity Scores
Description: The Low Back Pain Numeric Rating Scale (LBP NRS) is a standardized adaptation of the Pain Numeric Rating Scale for assessing pain intensity specifically related to the lower back. It uses an 11-point scale from 0 ("no low back pain") to 10 ("worst low back pain imaginable"), allowing patients to rate their pain over the past week.
Time Frame: Difference between the Day 1 (pre-intervention) and post-intervention at Week 4 (post-intervention - pre-intervention)
Population: individuals with chronic low back pain
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Number analyzed (Participants) | 26 | 25 | 20 | 22
score on a scale | -1.39 [-2.07 to -0.7] | -1.08 [-1.78 to -0.38] | -1.45 [-2.24 to -0.06] | -1.59 [-2.34 to -0.84]

3. Secondary Outcome: Cerebral Blood Flow (CBF) Differences Before and After Treatments
Description: Investigators will examine Cerebral blood flow (CBF) changes before and after treatment in several pain-related brain areas. Cerebral blood flow represents the volume of blood delivered to brain tissue per unit time, CBF data will be collected during arterial spin labeling (ASL) scans that will take place before the first treatment and after the last treatment. Images from these scans will be aggregated to an average CBF-weighted image to be used for analysis. In this report, we focused on bilateral postcentral Gyrus (MNI coordinate: +/-18, -34, 56, 2 mm sphere)
Time Frame: Day 1 (pre-intervention); post-intervention at Week 4
Population: chronic low back pain patients
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Number analyzed (Participants) | 20 | 19 | 18 | 17
mL/s | 3.3 (9.7) | -2.8 (9.6) | 2.7 (4.7) | 3.9 (17.9)

4. Secondary Outcome: Quantitative Sensory Testing (QST) Differences
Description: Participants' quantitative sensory testing (QST) ratings were analyzed before and after all treatments. Here, we report the heat pain threshold measured around the affected lower back area.
Time Frame: Day 1 (pre-intervention); post-intervention at Week 4 (pre-intervention - post-intervention)
Population: patients with chronic low back pain
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Number analyzed (Participants) | 25 | 22 | 19 | 20
degrees Celsius | -0.2 (2.2) | 1.0 (2.0) | -1 (1.7) | -0.6 (2)

5. Secondary Outcome: Primary Motor Cortex (M1) rsFC Changes Before and After 4-week Treatments
Description: We investigated whether tDCS and acupuncture treatments modulate resting-state functional connectivity (rsFC) of the M1. This was evaluated by comparing pre- and post-treatment MRI scans. In this report, we focused on the rsFC between the PAG and the rostral anterior cingulate cortex (rACC), using a seed defined by the rACC peak MNI coordinate (0, 34, 20) with a 2-mm radius sphere.
  Functional connectivity values were computed as Pearson's correlation coefficients between the mean time series of predefined regions of interest (ROIs). To improve normality and enable parametric statistical analysis, these correlation coefficients (r) were converted to Fisher z values using the transformation z = 0.5 × ln[(1 + r) / (1 - r)]. Higher Fisher z values indicate stronger positive connectivity, whereas lower values indicate weaker or negative connectivity. Changes in Fisher z values from baseline to post-intervention
Time Frame: Day 1 (pre-intervention); post-intervention at Week 4 (pre-intervention - post-intervention)
Population: low back pain patients
Measure: Mean (Standard Deviation); unit: Fisher z-transformed correlation coeffic
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
Number analyzed (Participants) | 24 | 23 | 19 | 21
Fisher z-transformed correlation coeffic | 0.14 (0.14) | -0.01 (0.18) | -0.03 (0.16) | 0 (0.13)

ADVERSE EVENTS:
Time Frame: from baseline to post-intervention assessments, up to 6 weeks
Description: Same as clinicaltrials.gov definition
Arm/Group | Verum Acupuncture + Real tDCS | Sham Acupuncture + Real tDCS | Verum Acupuncture + Sham tDCS | Sham Acupuncture + Sham tDCS
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/25 | 0/20 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/25 | 0/20 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 1/25 | 0/20 | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Verum Acupuncture + Real tDCS (N=27) | Sham Acupuncture + Real tDCS (N=25) | Verum Acupuncture + Sham tDCS (N=20) | Sham Acupuncture + Sham tDCS (N=23)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Some participants experienced headaches during and after the intervention, which resolved spontaneously without the need for additional treatment.
Needle pain discomfort (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — A participant reported residual needle discomfort after the intervention.
Neck pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — a participant reported neck pain that believed not related to this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03716830/Prot_SAP_000.pdf